CLINICAL TRIAL: NCT01707511
Title: Cohort Study on Patients Underwent Colorectal Surgery
Brief Title: The Investigation of the EtCO₂- PaCO₂ Relation During Laparoscopic Colon Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Ozmen, principal İnvestigator, Diskapi Teaching and Research Hospital
Other Study IDs: Diskapianesthesia-01
Record Dates: First submitted 2012-09-15; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Colorectal Cancer
Keywords: Arterial carbondioxide pressure; Colon surgery; End-tidal carbondioxide; Laparoscopic Trendelenburg
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Et-C02 is used to predict PaCO2 during surgery. There are controversies regarding the value of ETCO2 to predict PaCO2. The aim of this study was to investigate the relation between Et-CO₂ and PaCO₂ measurements in patients undergoing laparoscopic colorectal surgery. Patient and surgical characteristics, mechanical ventilation adjustments, and intraabdominal pressure values and the corelation between these parameters and EtCO₂ - PaCO₂ difference were also investigated.

DETAILED DESCRIPTION:
Patient records from patients underwent colorectal surgery between 2010-2011 will be studied. It was planned to include patients undergoing laparoscopic colorectal surgery with a predetermined anaesthesia protocol.

Patients will receive a standardized general anesthetic and thoracal epidural anaesthesia. Ventilatory parameters will be adjusted to maintain ETCO2 35 mmHg, Paw 25 cmH2O.Patient age, gen-der, BMI, ASA classification, the duration of surgery, anesthesia, Trendelenburg position and pneumoperitoneum. Hemodynamic parameters, blood gas analyzes, ventilation parameters and EtCO₂ values will be recorded. We determined 6 timelines to compare the difference between PaCO₂ and EtCO₂. These timelines were the times where we could collect the most data regarding blood gas analyzes. Preoperative period: to, 10th minute after the first insuflation and trendelendburg position: t₁,the first hour after the first insuflation and trendelendburg position: t₂, 10th minute after desuflation and supine position: t₃, 10th minute after the second insuflation and trendelendburg position: t₄, and 10th minute after the second desuflation and supine position:t₅. Primary outcome measure is the difference between PaCO₂ and EtCO₂ a difference greater than 5 mmHg was assumed to be important.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients underwent laparoscopic colorectal resection

Exclusion Criteria:

* convertion to the open surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled whom planned for elective laparoscopic colorectal resection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Ozmen, MD, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Teaching and Research Hospital, Ankara, Altindag, Turkey (Türkiye)